CLINICAL TRIAL: NCT05612607
Title: Switched Memory B-cells as a Marker for Humoral Immune System Recovery in Patients With Secondary Antibody Deficiency Due to Hematological Malignancies
Acronym: SAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20220516-01H
Record Dates: First submitted 2022-10-01; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Secondary Antibody Deficiency

STUDY DESIGN:
Intervention Model Description: Patients will be tested to determine SMB cell proportion/SMB cell levels for eligibility for IGRT discontinuation. If SMB cells are ≥ 2%, IGRT will be discontinued. If SMB cells are < 2%, the patient will remain on IGRT and a maximum of 40 mL of blood will be drawn again in 3-6 months to reassess SMB levels and eligibility for IGRT discontinuation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGRT discontinuation (Other): Participants will be tested to determine Switched memory B cells (SMB) levels. If SMB cells are ≥ 2%, IGRT will be discontinued. If SMB cells are < 2%, the patient will remain on IGRT and a maximum of 40 mL of blood will be drawn again in 3-6 months to reassess SMB levels and eligibility for IGRT discontinuation.
  Interventions: Drug: Immunoglobulin replacement therapy (IGRT)

INTERVENTIONS:
Drug: Immunoglobulin replacement therapy (IGRT) — IGRT discontinuation will be dependent on participant's SMB levels. If SMB cells are ≥ 2%, IGRT will be discontinued. If SMB cells are < 2%, the patient will remain on IGRT and a maximum of 40 mL of blood will be drawn again in 3-6 months to reassess SMB levels and eligibility for IGRT discontinuation.

SUMMARY:
Current treatment for patients with secondary antibody deficiency (SAD) is Immunoglobulin replacement therapy (IGRT). There are currently no clinical guidelines for IGRT discontinuation in patients with SAD. This study will examine the IGRT discontinuation success rate and IGRT discontinuation rate in patients.

DETAILED DESCRIPTION:
Immunoglobulin replacement therapy (IGRT) is a mainstay treatment for SAD and has been shown to reduce the risk of infection and increase quality of life in patients with SAD. Current guidelines recommend that patients with severe hypogammaglobulinemia (IgG <4 g/L) or patients with a history of recurrent or severe infections should be offered IGRT, which can be administered intravenously on a monthly basis or more frequently by subcutaneous infusions. There are currently no clinical guidelines for IGRT discontinuation. Although research conducted at the Ottawa Hospital indicates successful discontinuation of IGRT, clinicians need a tool to predict the recovery of humoral immunity and the risk of infection in these patients in order to determine whether IGRT may be safely discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. History of leukemia, lymphoma, or plasma cell disease
2. Receiving IGRT for SAD for at least 12 months
3. Over 18 years of age
4. Able to provide informed consent
5. Able to speak English or French
6. Available for ongoing follow-up as required

Exclusion Criteria:

1. Receiving chemotherapy or immune-oncology treatment during the study period
2. Severe infection within the last 6 months
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
IGRT discontinuation sucess rate | 12 months post discontinuation
  IGRT discontinuation success rate defined as the proportion of patients with normal SMB levels who stop IGRT and experience less than or equal to 1 moderate infection and no severe infection within 12 months of IGRT discontinuation. Moderate infection will be defined as an infection that requires outpatient oral antimicrobial treatment. Severe infection will be defined as an infection that requires intravenous antimicrobial treatment and/or hospitalization.
IGRT discontinuation rate | 12 months post discontinuation
  IGRT discontinuation rate defined as the proportion of recruited adult patients with SAD who discontinue IGRT during the study period.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life | Through study completion, an average of 1 year
  Change in Health-Related Quality of Life (HRQoL) before and after IGRT discontinuation. The 36-item Short Form Survey (SF-36, RAND Corporation) will be used to obtain HRQoL data.
Change in Health-Related Quality of Life | Through study completion, an average of 1 year
  Change in Health-Related Quality of Life (HRQoL) before and after IGRT discontinuation. The Euroqol 5-dimension 5-level (EQ-5D-5L) questionnaire will be used to obtain HRQoL data.
Cost saving potential | Through study completion, an average of 1 year
  Calculated potential cost saving based on the study IGRT discontinuation rate using SMB as a marker for discontinuation.
Receiver operating curve (ROC) | Through study completion, an average of 1 year
  We will estimate a receiver operating curve (ROC) of SMB proportion as a predictor of successful discontinuation.